CLINICAL TRIAL: NCT01209325
Title: AMC-072: Protective Effect of Quadrivalent Vaccine in Young HIV-Positive Males Who Have Sex With Males
Brief Title: Vaccine Therapy in Preventing Human Papillomavirus Infection in Young HIV-Positive Male Patients Who Have Sex With Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other); Merck Sharp & Dohme LLC (Industry); AIDS and Cancer Specimen Resource (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMC-072; AMC-072 (Other: AMC); U01CA121947 (NIH); CDR0000685816 (Other: NCI)
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Anal Cancer; Nonneoplastic Condition; Penile Cancer; Precancerous Condition
Keywords: human papilloma virus infection; anal cancer; penile cancer; HIV infection
MeSH Terms: conditions — Anus Neoplasms; Penile Neoplasms; Precancerous Conditions; Papillomavirus Infections; HIV Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccination (Experimental): Gardasil (quadrivalent HPV types 6, 11, 16, 18) vaccination at weeks 0, 8, 24.
  Interventions: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus may help the body build an effective immune response to prevent viral infection.

PURPOSE: This phase II trial is studying how well vaccine therapy works in preventing human papillomavirus (HPV) infection in young HIV-positive male patients who have sex with males.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the protective effect of the HPV-6, -11, -16, -18 vaccine in preventing penile/scrotal condyloma and HPV-6, -11, -16, -18- associated perianal/anal disease in HIV-positive males who have sex with males (MSM) age 13-26 years by comparing the incidence of these lesions among those naïve to the relevant HPV type(s) at baseline to those who are not naïve at baseline.
* To determine the protective effect of the HPV-6, -11, -16, -18 vaccine in preventing persistent anogenital infection with HPV-6, -11, -16, or 18 in HIV-positive MSM age 13-26 years by comparing the incidence of persistent infection among those naïve to the relevant HPV type(s) at baseline to those who are not naïve at baseline.
* To determine the protective effect of the HPV-6, -11, -16, -18 vaccine in preventing anogenital lesions associated with HPV 6,-11,-16, -18 and persistent infection with these types, in HIV-positive MSM age 13-26 years by comparing the incidence of lesions and persistent infection among those naïve to the relevant types at baseline to incident lesions and infection among MSM naïve to these HPV types who participated in the Merck 020 protocol and who received placebo as part of the protocol.

Secondary

* To define the safety of the HPV-6, -11, -16, -18 vaccine in HIV-positive MSM age 13-26 years.
* To evaluate the levels and persistence of HPV 6, 11, 16 and 18 Ab titers after the vaccination series among subjects who are seropositive and seronegative at baseline.
* To examine whether the protective effect and antibody titers vary as a function of the following at the time of initial vaccination: subject age, HAART treatment status, HIV viral load, CD4 + T-cell count, and nadir CD4 level.

Tertiary

* To quantify anogenital HPV DNA viral load prior to and after receipt of the quadrivalent HPV vaccine.
* To identify and quantify HPV types in the oral cavity of HIV-positive MSM prior to and after receipt of the quadrivalent HPV vaccine.
* To identify HPV strain variants among HIV-positive participants prior to and after receipt of the quadrivalent HPV vaccine.
* Assess the prevalence and incidence of urinary and gonorrhea and Chlamydia trachomatis infection at baseline and their relationship with prevalent and incident anogenital HPV infection and anal condyloma or AIN.
* To characterize young men's risk perceptions, sexual behaviors, and STI diagnosis after HPV vaccination.

OUTLINE: This is a multicenter study.

Patients receive quadrivalent human papillomavirus (types 6, 11, 16, and 18) recombinant vaccine intramuscularly on day 1 and in weeks 8 and 24.

Blood and tissue samples may be collected periodically for laboratory studies.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Men with a history of at least one male sexual partner

  * "Men" is defined as those documented "male" at birth (including male-to-female transgendered persons)
* HIV-1 infection as documented by any federally approved, licensed HIV test performed in conjunction with screening (ELISA, western blot, or other approved test)

  * Alternatively, this documentation may include a record that another physician has documented that the patient has HIV based on prior ELISA and western blot, or other approved diagnostic tests
* Meets one of the following sets of criteria:

  * Patients receiving antiretroviral therapy:

    * Receipt of antiretroviral therapy for at least 3 months prior to entry
    * No change in antiretroviral therapy within 30 days prior to entry
  * Patients not receiving antiretroviral therapy:

    * CD4-cell count ≥ 350 cells/mm³ within 90 days prior to study entry
    * No plans to start antiretroviral therapy prior to Week 28
* Normal anal cytological result, LSIL/condyloma, or ASCUS result within 90 days prior to entry, and no HGAIN on biopsy

  * No current or history of anal or peri-anal carcinoma
  * No anal cytological result of HSIL, atypical squamous cells suggestive of HSIL (ASC-H), or suggestive of invasive carcinoma at screening; or history of these results
* No presence of penile or scrotal condyloma, LGAIN (condyloma or AIN 1), HGAIN (e.g., AIN 2 or 3, or perianal intraepithelial neoplasia grade 2 or 3), or invasive carcinoma at pre-entry on biopsy
* No history of HGAIN

PATIENT CHARACTERISTICS:

* Karnofsky performance score ≥ 70 within 45 days prior to entry
* Absolute neutrophil count (ANC) > 750 cells/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* AST (SGOT), ALT (SGPT) ≤ 3 times upper limit of normal (ULN)
* Total or conjugated (direct) bilirubin ≤ 2.5 times ULN within 45 days before study entry, with the exception of isolated hyperbilirubinemia that is considered due to atazanavir
* Calculated creatinine clearance ≥ 60 mL/min
* No hemophilia
* No active drug or alcohol use or dependence that, in the opinion of the site Investigator, would interfere with adherence to study requirements
* No serious illness requiring systemic treatment and/or hospitalization within 45 days prior to entry
* No serious medical or psychiatric illness that, in the opinion of the site Investigator, will interfere with the ability of the subject to give informed consent or adhere to the protocol
* No allergy to yeast or any of the components of Gardasil

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior splenectomy
* No prior receipt of Gardasil or other HPV vaccine
* No use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids for greater than 14 days, investigational vaccines, interleukins, interferons, growth factors, or IVIG within 45 days prior to study entry
* No expected use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids used for greater than 14 days, investigational vaccines, interleukins, interferons, growth factors, or IVIG during study followup

  * No patients with hepatitis C who expect to initiate treatment for hepatitis C (e.g., interferons) during this trial
* Not currently receiving anticoagulation therapy other than acetylsalicylic acid

Ages: 13 Years to 26 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 149 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Principal Investigator — University of California, San Francisco
Locations (18):
- United States (17):
  - Moores UCSD Cancer Center, La Jolla, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Ruth M. Rothstein Core Center at Cook County Hospital, Chicago, Illinois
  - Fenway Community Health, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Laser Surgery Care, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - St. Jude's Children's Research Hospital, Memphis, Tennessee
  - Thomas Street Health Center, Houston, Texas
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- University of Puerto Rico Comprehensive Cancer Center, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahn JA, Belzer M, Chi X, Lee J, Gaur AH, Mayer K, Martinez J, Futterman DC, Stier EA, Paul ME, Chiao EY, Reirden D, Goldstone SE, Ortiz Martinez AP, Cachay ER, Barroso LF, Da Costa M, Wilson CM, Palefsky JM; AIDS Malignancy Consortium and Adolescent Medicine Trials Network for HIV/AIDS Interventions. Pre-vaccination prevalence of anogenital and oral human papillomavirus in young HIV-infected men who have sex with men. Papillomavirus Res. 2019 Jun;7:52-61. doi: 10.1016/j.pvr.2019.01.002. Epub 2019 Jan 15. PMID 30658128

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccination: Gardasil (quadrivalent HPV types 6, 11, 16, 18) vaccination at weeks 0, 8, 24.
  quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine
  laboratory biomarker analysis
Period: Overall Study
Arm/Group | Vaccination
Started (Enrolled) | 149
Eligible | 145
Received First Vaccine Injection | 144
Received Second Vaccine Injection | 141
Received Third Vaccine Infjection | 138
Returned After Week 28 | 124
Completed | 106
Not Completed | 43
Not completed — Lost to Follow-up | 24
Not completed — Adverse Event | 1
Not completed — Relocated | 3
Not completed — Refusal after starting therapy | 8
Not completed — Protocol Violation | 4
Not completed — Refusal prior to therapy | 1
Not completed — Incarceration | 2

BASELINE CHARACTERISTICS:
Population: Eligible participants who received at least one dose of vaccine.
Arm/Group | Vaccination
Number analyzed (Participants) | 144
Age, Continuous [Mean (Full Range); unit: years] | 23.5 [18.1 to 27.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 80
  White | 46
  More than one race | 3
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 3
  United States | 141

OUTCOME MEASURES:

1. Primary Outcome: Incidence of AIN or Anal/Perianal Condyloma Associated With HPV 6 DNA
Description: Incident events are defined as having AIN (e.g., AIN or anal/perianal condyloma) with HPV 6 positive DNA in participants without HPV-6 related AIN at baseline.
Time Frame: Post Month 7 through Month 24
Population: Eligible participants without prevalent HPV 6 related AIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: Events per 100 person years
Groups:
- Naive to HPV 6: HPV 6 negative based on serum at visit 0 and DNA from visit 0 and 3 from any anatomical site.
- Prior Exposure to HPV 6: HPV 6 positive based on serum at visit 0.
Arm/Group | Naive to HPV 6 | Prior Exposure to HPV 6
Number analyzed (Participants) | 15 | 34
Events per 100 person years | 0.0 | 11.1
Statistical Analysis 1: Comparison: Naive to HPV 6 vs Prior Exposure to HPV 6; Test type: Superiority; p = 0.112, Exact poisson test — Two-sided p-value
Statistical Analysis 2: Comparison: Naive to HPV 6; This study's Naive to HPV 6 group was compared to the per-protocol Merck 020 historical placebo group naive to HPV 6 (NCT00090285), 0.0 events per 100 person years (PY) versus 3.4 events per 100 PY, respectively; Test type: Superiority; p = 0.447, Exact Poisson calculation — One-sided test

2. Primary Outcome: Incidence of AIN or Anal/Perianal Condyloma Associated With HPV 11 DNA
Description: Incident events are defined as having AIN (e.g., AIN or anal/perianal condyloma) with HPV 11 positive DNA in participants without HPV-11 related AIN at baseline.
Time Frame: Post Month 7 through Month 24
Population: Eligible participants without prevalent HPV 11 related AIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: Events per 100 person years
Groups:
- Naive to HPV 11: HPV 11 negative based on serum at visit 0 and DNA from visit 0 and 3 from any anatomical site.
- Prior Exposure to HPV 11: HPV 11 positive based on serum at visit 0.
Arm/Group | Naive to HPV 11 | Prior Exposure to HPV 11
Number analyzed (Participants) | 35 | 28
Events per 100 person years | 0.0 | 2.2
Statistical Analysis 1: Comparison: Naive to HPV 11 vs Prior Exposure to HPV 11; Test type: Superiority; p = 0.224, Exact poisson test — Two-sided p-value
Statistical Analysis 2: Comparison: Naive to HPV 11; This study's Naive to HPV 11 group was compared to the per-protocol Merck 020 historical placebo group naive to HPV 11 (NCT00090285), 0.0 events per 100 person years (PY) versus 2.0 events per 100 PY, respectively; Test type: Superiority — One-sided p-value; p = 0.361, Exact Poisson calculation

3. Primary Outcome: Incidence of AIN or Anal/Perianal Condyloma Associated With HPV 16 DNA
Description: Incident events are defined as having AIN (e.g., AIN or anal/perianal condyloma) with HPV 16 positive DNA in participants without HPV-16 related AIN at baseline.
Time Frame: Post Month 7 through Month 24
Population: Eligible participants without prevalent HPV 16 related AIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: Events per 100 person years
Groups:
- Naive to HPV 16: HPV 16 negative based on serum at visit 0 and DNA from visit 0 and 3 from any anatomical site.
- Prior Exposure to HPV 16: HPV 16 positive based on serum at visit 0.
Arm/Group | Naive to HPV 16 | Prior Exposure to HPV 16
Number analyzed (Participants) | 39 | 29
Events per 100 person years | 0.0 | 4.5
Statistical Analysis 1: Comparison: Naive to HPV 16 vs Prior Exposure to HPV 16; Test type: Superiority; p = 0.079, Exact poisson test — Two-sided p-value
Statistical Analysis 2: Comparison: Naive to HPV 16; This study's Naive to HPV 16 group was compared to the per-protocol Merck 020 historical placebo group naive to HPV 16 (NCT00090285), 0.0 events per 100 person years (PY) versus 1.8 events per 100 PY, respectively; Test type: Superiority; p = 0.350, Exact Poisson calculation — One-sided p-value

4. Primary Outcome: Incidence of AIN or Anal/Perianal Condyloma Associated With HPV 18 DNA
Description: Incident events are defined as having AIN (e.g., AIN or anal/perianal condyloma) with HPV 18 positive DNA in participants without HPV-18 related AIN at baseline.
Time Frame: Post Month 7 through Month 24
Population: Eligible participants without prevalent HPV 18 related AIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: Events per 100 person years
Groups:
- Naive to HPV 18: HPV 18 negative based on serum at visit 0 and DNA from visit 0 and 3 from any anatomical site.
- Prior Exposure to HPV 18: HPV 18 positive based on serum at visit 0.
Arm/Group | Naive to HPV 18 | Prior Exposure to HPV 18
Number analyzed (Participants) | 47 | 23
Events per 100 person years | 0.0 | 2.8
Statistical Analysis 1: Comparison: Naive to HPV 18 vs Prior Exposure to HPV 18; Test type: Superiority; p = 0.162, Exact poisson test
Statistical Analysis 2: Comparison: Naive to HPV 18; This study's Naive to HPV 18 group was compared to the Merck 020 per-protocol historical placebo group naive to HPV 18 (NCT00090285), 0.0 events per 100 person years (PY) versus 1.0 events per 100 PY, respectively; Test type: Superiority; p = 0.490, Exact Poisson calculation — One-sided p-value

5. Primary Outcome: Incidence of Persistent Anogenital Infection With HPV 6 DNA
Description: Incident events are defined as having HPV 6 positive PCR results at 2 or more consecutive visits in those who were DNA negative for HPV 6. Persistence was defined based on being persistent in the same anatomical site.
Time Frame: Post Month 7 through Month 24
Population: All eligible participants who were HPV 6 DNA negative at baseline and received at least one vaccination and returned after month 7 with evaluable PCR tests at two consecutive visits.
Measure: Number; unit: events per 100 person years
Groups:
- Prior Exposure HPV 6: HPV 6 positive based on serum at visit 0 from any anatomical site.
Arm/Group | Naive to HPV 6 | Prior Exposure HPV 6
Number analyzed (Participants) | 29 | 15
events per 100 person years | 1.8 | 0.0
Statistical Analysis 1: Comparison: Naive to HPV 6 vs Prior Exposure HPV 6; Test type: Superiority; p = 0.671, Exact Poisson calculation — Two-sided p-value is comparing naive and prior exposure groups for HPV 6
Statistical Analysis 2: Comparison: Naive to HPV 6; This study's Naive to HPV 6 group was compared to the per-protocol Merck 020 historical placebo group naive to HPV 6 (NCT00090285), 1.8 events per 100 person years (PY) versus 4.5 events per 100 PY, respectively; Test type: Superiority; p = 0.312, Exact Poisson calculation — One-sided p-value

6. Primary Outcome: Incidence of Persistent Anogenital Infection With HPV 11 DNA
Description: Incident events are defined as having positive PCR results with HPV 11 at 2 or more consecutive visits in those who were DNA negative for HPV 11 at baseline. Persistence was defined based on being persistent in the same anatomical site.
Time Frame: Post Month 7 through Month 24
Population: All eligible participants who were HPV 11 DNA negative at baseline and received at least one vaccination and returned after month 7 with evaluable PCR tests at two consecutive visits.
Measure: Number; unit: events per 100 person years
Groups:
- Prior Exposure to HPV 11: HPV 11 positive based on serum at visit 0 from any anatomical site.
Arm/Group | Naive to HPV 11 | Prior Exposure to HPV 11
Number analyzed (Participants) | 55 | 33
events per 100 person years | 0.0 | 0.0
Statistical Analysis 1: Comparison: Naive to HPV 11 vs Prior Exposure to HPV 11; Test type: Superiority; p > 0.999, Exact Poisson calculation — Two-sided p-value
Statistical Analysis 2: Comparison: Naive to HPV 11; This study's Naive to HPV 11 group was compared to the per-protocol Merck 020 historical placebo group naive to HPV 11 (NCT00090285), 0.0 events per 100 person years (PY) versus 1.7 events per 100 PY, respectively; Test type: Superiority; p = 0.209, Exact Poisson calculation — One-sided p-value

7. Primary Outcome: Incidence of Persistent Anogenital Infection With HPV 16 DNA
Description: Incident events are defined as having positive PCR results with HPV 16 at 2 or more consecutive visits in those who were DNA negative for HPV 16 at baseline. Persistence was defined based on being persistent in the same anatomical site.
Time Frame: Post Month 7 through Month 24
Population: All eligible participants who were HPV 16 DNA negative at baseline and received at least one vaccination and returned after month 7 with evaluable PCR tests at two consecutive visits.
Measure: Number; unit: events per 100 person years
Groups:
- Prior Exposure to HPV 16: HPV 16 positive based on serum at visit 0 from any anatomical site.
Arm/Group | Naive to HPV 16 | Prior Exposure to HPV 16
Number analyzed (Participants) | 54 | 23
events per 100 person years | 2.9 | 0.0
Statistical Analysis 1: Comparison: Naive to HPV 16 vs Prior Exposure to HPV 16; Test type: Superiority; p = 0.386, Exact Poisson calculation — Two-sided p-value
Statistical Analysis 2: Comparison: Naive to HPV 16; This study's Naive to HPV 16 group was compared to the per-protocol Merck 020 historical placebo group naive to HPV 16 (NCT00090285), 2.9 events per 100 person years (PY) versus 4.9 events per 100 PY, respectively; Test type: Superiority; p = 0.305, Exact Poisson calculation — One-sided test

8. Primary Outcome: Incidence of Persistent Anogenital Infection With HPV 18 DNA
Description: Incident events are defined as having positive PCR results with HPV 18 at 2 or more consecutive visits in those who were DNA negative for HPV 18. Persistence was defined based on being persistent in the same anatomical site.
Time Frame: Post Month 7 through Month 24
Population: All eligible participants who were HPV 18 DNA negative at baseline and received at least one vaccination and returned after month 7 with evaluable PCR tests at two consecutive visits.
Measure: Number; unit: events per 100 person years
Groups:
- Prior Exposure to HPV 18: HPV 18 positive based on serum at visit 0 from any anatomical site.
Arm/Group | Naive to HPV 18 | Prior Exposure to HPV 18
Number analyzed (Participants) | 74 | 23
events per 100 person years | 0.7 | 0.0
Statistical Analysis 1: Comparison: Naive to HPV 18; Test type: Superiority; p = 0.622, Exact Poisson calculation — Two-sided p-value
Statistical Analysis 2: Comparison: Naive to HPV 18; This study's Naive to HPV 18 group was compared to the per-protocol Merck 020 historical placebo group naive to HPV 18 (NCT00090285), 0.7 events per 100 person years (PY) versus 2.7 events per 100 PY, respectively; Test type: Superiority; p = 0.150, Exact Poisson calculation — One-sided p-value

9. Primary Outcome: Incidence of HGAIN Associated With HPV 6
Description: Incident events are defined as having HGAIN (e.g., AIN 2 or 3, or perianal intraepithelial neoplasia grade 2 or 3) with HPV 6 positive DNA in participants without HPV 6 related HGAIN at baseline.
Time Frame: Post month 7 through month 24
Population: Eligible participants without prevalent HPV 6 related HGAIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 6 | Prior Exposure to HPV 6
Number analyzed (Participants) | 15 | 56
per 100 person years | 0.0 | 10.4
Statistical Analysis 1: Comparison: Naive to HPV 6 vs Prior Exposure to HPV 6; Test type: Superiority; p = 0.064, Exact Poisson calculation — Two-sided p-value

10. Primary Outcome: Incidence of HGAIN Associated With HPV 11
Description: Incident events are defined as having HGAIN (e.g., AIN 2 or 3, or perianal intraepithelial neoplasia grade 2 or 3) with HPV 11 positive DNA in participants without HPV 11 related HGAIN at baseline.
Time Frame: Post month 7 through month 24
Population: Eligible participants without prevalent HPV 11 related HGAIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 11 | Prior Exposure to HPV 11
Number analyzed (Participants) | 35 | 36
per 100 person years | 0.0 | 1.7
Statistical Analysis 1: Comparison: Naive to HPV 11 vs Prior Exposure to HPV 11; Test type: Superiority; p = 0.745, Exact Poisson calculation — Two-sided test

11. Primary Outcome: Incidence of HGAIN Associated With HPV 16
Description: Incident events are defined as having HGAIN (e.g., AIN 2 or 3, or perianal intraepithelial neoplasia grade 2 or 3) with HPV 16 positive DNA in participants without HPV 16 related HGAIN at baseline.
Time Frame: Post month 7 through month 24
Population: Eligible participants without prevalent HPV 16 related HGAIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 16 | Prior Exposure to HPV 16
Number analyzed (Participants) | 39 | 32
per 100 person years | 0.0 | 8.4
Statistical Analysis 1: Comparison: Naive to HPV 16 vs Prior Exposure to HPV 16; Test type: Superiority; p = 0.014, Exact Poisson calculation

12. Primary Outcome: Incidence of HGAIN Associated With HPV 18
Description: Incident events are defined as having HGAIN (e.g., AIN 2 or 3, or perianal intraepithelial neoplasia grade 2 or 3) with HPV 18 positive DNA in participants without HPV 18 related HGAIN at baseline.
Time Frame: Post month 7 through month 24
Population: Eligible participants without prevalent HPV 18 related HGAIN at baseline who received at least one vaccination and returned after month 7 with evaluable anal/perianal histology and PCR samples.
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 18 | Prior Exposure to HPV 18
Number analyzed (Participants) | 47 | 24
per 100 person years | 0.0 | 2.7
Statistical Analysis 1: Comparison: Naive to HPV 18 vs Prior Exposure to HPV 18; Test type: Superiority; p = 0.166, Exact Poisson calculation — Two-sided p-value

13. Primary Outcome: Incidence of Penile/Scrotal Condyloma in HPV 6 Naive and Prior Exposed Participants
Description: Incident events are defined as having penile/scrotal warts reported clinically in participants penile/scrotal condyloma at baseline.
Time Frame: Post month 7 through month 24
Population: Eligible participants without penile/scrotal condyloma at baseline who received at least one vaccination and returned after month 7 with evaluable clinical assessments.
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 6 | Prior Exposure to HPV 6
Number analyzed (Participants) | 29 | 91
per 100 person years | 1.8 | 1.1
Statistical Analysis 1: Comparison: Naive to HPV 6 vs Prior Exposure to HPV 6; Test type: Superiority; p = 0.789, Exact Poisson calculation — Two-sided p-value

14. Primary Outcome: Incidence of Penile/Scrotal Condyloma in HPV 11 Naive and Prior Exposed Participants
Description: as for outcome 13
Time Frame: Post month 7 through month 24
Population: as for outcome 13
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 11 | Prior Exposure to HPV 11
Number analyzed (Participants) | 58 | 61
per 100 person years | 0.9 | 1.7
Statistical Analysis 1: Comparison: Naive to HPV 11 vs Prior Exposure to HPV 11; Test type: Superiority; p = 0.809, 0.809 — Two-sided p-value

15. Primary Outcome: Incidence of Penile/Scrotal Condyloma in HPV 16 Naive and Prior Exposed Participants
Description: as for outcome 13
Time Frame: Post month 7 through month 24
Population: as for outcome 13
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 16 | Prior Exposure to HPV 16
Number analyzed (Participants) | 56 | 63
per 100 person years | 1.8 | 0.8
Statistical Analysis 1: Comparison: Naive to HPV 16 vs Prior Exposure to HPV 16; Test type: Superiority; p = 0.422, Exact Poisson calculation — Two-sided p-value

16. Primary Outcome: Incidence of Penile/Scrotal Condyloma in HPV 18 Naive and Prior Exposed Participants
Description: as for outcome 13
Time Frame: Post month 7 through month 24
Population: as for outcome 13
Measure: Number; unit: per 100 person years
Arm/Group | Naive to HPV 18 | Prior Exposure to HPV 18
Number analyzed (Participants) | 76 | 44
per 100 person years | 0.7 | 2.3
Statistical Analysis 1: Comparison: Naive to HPV 18 vs Prior Exposure to HPV 18; Test type: Superiority; p = 0.423, Exact Poisson calculation — Two-sided p-value

17. Secondary Outcome: Occurrence of Grade ≥ 3 Adverse Events (AEs) That Were Possibly, Probably, or Definitely Related to the Vaccine
Description: Number of participants who experienced grade 3 and higher AEs that were possibly, probably or definitely related to the vaccine.
Time Frame: Through Month 24
Population: The safety population included eligible participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination
Number analyzed (Participants) | 144
Participants | 0

18. Secondary Outcome: Geometric Mean Titers for HPV 6
Description: Geometric mean concentration of antibodies for HPV 6 at each visit
Time Frame: Baseline through month 24
Population: Eligible participants who received at least one vaccination with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- HPV 6 Sero-negative at Baseline: Sero-negative for HPV 6 at baseline.
- HPV 6 Sero-positive at Baseline: Sero-positive for HPV 6 at baseline
Arm/Group | HPV 6 Sero-negative at Baseline | HPV 6 Sero-positive at Baseline
Number analyzed (Participants) | 50 | 93
mMU/mL
  Baseline | 0 [0 to 0] | 81.7 [64.5 to 851.8]
  Month 7: number analyzed (Participants) | 46 | 81
  Month 7 | 302.3 [236.4 to 386.6] | 637.8 [477.6 to 851.8]
  Month 12: number analyzed (Participants) | 43 | 75
  Month 12 | 111.8 [83.6 to 149.4] | 420.9 [318.2 to 556.7]
  Month 18: number analyzed (Participants) | 40 | 71
  Month 18 | 79.7 [55.8 to 113.9] | 335.3 [262.8 to 428.0]
  Month 24: number analyzed (Participants) | 38 | 66
  Month 24 | 73.7 [48.5 to 112.0] | 356.6 [272.4 to 466.8]

19. Secondary Outcome: Geometric Mean Titers for HPV 11
Description: Geometric mean concentration of antibodies for HPV 11 at each visit
Time Frame: Baseline through month 24
Population: Eligible participants who received at least one vaccination with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- HPV 11 Sero-negative at Baseline: Sero-negative for HPV 11 at baseline.
- HPV 11 Sero-positive at Baseline: Sero-positive for HPV 11 at baseline
Arm/Group | HPV 11 Sero-negative at Baseline | HPV 11 Sero-positive at Baseline
Number analyzed (Participants) | 79 | 64
mMU/mL
  Baseline | 0 [0 to 0] | 42.7 [30.1 to 60.5]
  Month 7: number analyzed (Participants) | 71 | 56
  Month 7 | 452.4 [378.1 to 541.4] | 976.2 [757.5 to 1258.1]
  Month 12: number analyzed (Participants) | 67 | 51
  Month 12 | 132.0 [102.7 to 169.8] | 493.7 [355.2 to 686.1]
  Month 18: number analyzed (Participants) | 63 | 48
  Month 18 | 89.6 [67.2 to 119.4] | 373.2 [262.1 to 531.6]
  Month 24: number analyzed (Participants) | 60 | 44
  Month 24 | 84.4 [62.1 to 114.9] | 300.2 [205.8 to 438.1]

20. Secondary Outcome: Geometric Mean Titers for HPV 16
Description: Geometric mean concentration of antibodies for HPV 16 at each visit
Time Frame: Baseline through 24 months
Population: Eligible participants who received at least one vaccination with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- HPV 16 Sero-negative at Baseline: Sero-negative for HPV 16 at baseline.
- HPV 16 Sero-positive at Baseline: Sero-positive for HPV 16 at baseline
Arm/Group | HPV 16 Sero-negative at Baseline | HPV 16 Sero-positive at Baseline
Number analyzed (Participants) | 92 | 51
mMU/mL
  Baseline | 0 [0 to 0] | 66.6 [46.7 to 95.1]
  Month 7: number analyzed (Participants) | 82 | 45
  Month 7 | 1535.6 [1272.5 to 1853.1] | 2947.8 [2249.0 to 3863.6]
  Month 12: number analyzed (Participants) | 76 | 42
  Month 12 | 451.6 [352.5 to 578.5] | 1436.6 [1095.2 to 1884.6]
  Month 18: number analyzed (Participants) | 73 | 38
  Month 18 | 309.5 [237.6 to 403.1] | 1242.9 [892.2 to 1731.5]
  Month 24: number analyzed (Participants) | 67 | 37
  Month 24 | 272.4 [195.5 to 379.6] | 1079.5 [771.8 to 1510.0]

21. Secondary Outcome: Geometric Mean Titers for HPV 18
Description: Geometric mean concentration of antibodies for HPV 18 at each visit
Time Frame: Baseline through 24 months
Population: Eligible participants who received at least one vaccination with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- HPV 18 Sero-negative at Baseline: Sero-negative for HPV 18 at baseline.
- HPV 18 Sero-positive at Baseline: Sero-positive for HPV 18 at baseline
Arm/Group | HPV 18 Sero-negative at Baseline | HPV 18 Sero-positive at Baseline
Number analyzed (Participants) | 104 | 39
mMU/mL
  Baseline | 0 [0 to 0] | 41.3 [28.1 to 60.7]
  Month 7: number analyzed (Participants) | 94 | 33
  Month 7 | 294.2 [232.8 to 371.8] | 482.2 [351.9 to 660.7]
  Month 12: number analyzed (Participants) | 88 | 30
  Month 12 | 63.1 [48.7 to 81.6] | 214.6 [141.0 to 326.6]
  Month 18: number analyzed (Participants) | 82 | 29
  Month 18 | 39.2 [29.7 to 51.7] | 244.3 [158.0 to 377.5]
  Month 24: number analyzed (Participants) | 73 | 31
  Month 24 | 39.0 [28.7 to 52.8] | 161.9 [103.3 to 253.7]

22. Secondary Outcome: Geometric Mean Titers for HPV 6 According to Participant Age, HIV Viral Load, CD4+ T Cell Count, and Nadir CD4 Level
Description: Geometric mean concentration of antibodies for HPV 6 at 7 and 24 months
Time Frame: at 7 and 24 Months
Population: Eligible participants who received at least one vaccination and who were sero-negative for HPV 6 at baseline with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Month 7 Visit: Month 7 visit after enrollment
- Month 24 Visit: Month 24 visit after enrollment
Arm/Group | Month 7 Visit | Month 24 Visit
Number analyzed (Participants) | 43 | 38
mMU/mL
  Age<24 years: number analyzed (Participants) | 24 | 22
  Age<24 years | 319 [227 to 451] | 71 [42 to 121]
  Age>=24 years: number analyzed (Participants) | 19 | 16
  Age>=24 years | 304 [200 to 463] | 77 [37 to 163]
  Baseline HIV viral load <=75: number analyzed (Participants) | 37 | 32
  Baseline HIV viral load <=75 | 324 [244 to 431] | 81 [53 to 125]
  Baseline HIV viral load >75: number analyzed (Participants) | 6 | 6
  Baseline HIV viral load >75 | 250 [118 to 528] | 45 [8 to 257]
  Baseline CD4 <=500: number analyzed (Participants) | 12 | 11
  Baseline CD4 <=500 | 341 [178 to 657] | 97 [44 to 212]
  Baseline CD4 >500: number analyzed (Participants) | 31 | 27
  Baseline CD4 >500 | 302 [229 to 399] | 66 [39 to 111]
  Nadir CD4 <=350: number analyzed (Participants) | 17 | 16
  Nadir CD4 <=350 | 361 [222 to 584] | 77 [38 to 155]
  Nadir CD4>350: number analyzed (Participants) | 23 | 21
  Nadir CD4>350 | 300 [214 to 421] | 75 [42 to 134]

23. Secondary Outcome: Geometric Mean Titers for HPV 11 According to Participant Age, HIV Viral Load, CD4+ T Cell Count, and Nadir CD4 Level
Description: Geometric mean concentration of antibodies for HPV 11 at 7 and 24 months
Time Frame: at 7 and 24 Months
Population: Eligible participants who received at least one vaccination and who were sero-negative for HPV 11 at baseline with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Month 7 Visit | Month 24 Visit
Number analyzed (Participants) | 68 | 60
mMU/mL
  Age<24 years: number analyzed (Participants) | 37 | 33
  Age<24 years | 434 [336 to 561] | 71 [49 to 105]
  Age>=24 years: number analyzed (Participants) | 31 | 27
  Age>=24 years | 482 [361 to 645] | 104 [61 to 174]
  Baseline HIV viral load <=75: number analyzed (Participants) | 58 | 51
  Baseline HIV viral load <=75 | 473 [385 to 583] | 86 [63 to 118]
  Baseline HIV viral load >75: number analyzed (Participants) | 10 | 9
  Baseline HIV viral load >75 | 365 [226 to 587] | 75 [21 to 260]
  Baseline CD4 <=500: number analyzed (Participants) | 24 | 20
  Baseline CD4 <=500 | 475 [354 to 638] | 98 [59 to 163]
  Baseline CD4 >500: number analyzed (Participants) | 44 | 40
  Baseline CD4 >500 | 445 [347 to 571] | 78 [53 to 117]
  Nadir CD4 <=350: number analyzed (Participants) | 33 | 31
  Nadir CD4 <=350 | 469 [351 to 626] | 87 [57 to 133]
  Nadir CD4>350: number analyzed (Participants) | 32 | 28
  Nadir CD4>350 | 452 [344 to 594] | 82 [50 to 134]

24. Secondary Outcome: Geometric Mean Titers for HPV 16 According to Participant Age, HIV Viral Load, CD4+ T Cell Count, and Nadir CD4 Level
Description: Geometric mean concentration of antibodies for HPV 16 at 7 and 24 months
Time Frame: at 7 and 24 Months
Population: Eligible participants who received at least one vaccination and who were sero-negative for HPV 16 at baseline with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Month 7 Visit | Month 24 Visit
Number analyzed (Participants) | 76 | 66
mMU/mL
  Age<24 years: number analyzed (Participants) | 49 | 44
  Age<24 years | 1572 [1239 to 1995] | 268 [185 to 388]
  Age>=24 years: number analyzed (Participants) | 27 | 22
  Age>=24 years | 1467 [1013 to 2126] | 272 [131 to 566]
  Baseline HIV viral load <=75: number analyzed (Participants) | 68 | 57
  Baseline HIV viral load <=75 | 1630 [1328 to 2002] | 282 [200 to 398]
  Baseline HIV viral load >75: number analyzed (Participants) | 8 | 9
  Baseline HIV viral load >75 | 914 [441 to 1894] | 201 [51 to 795]
  Baseline CD4 <=500: number analyzed (Participants) | 27 | 24
  Baseline CD4 <=500 | 1556 [1123 to 2156] | 359 [218 to 590]
  Baseline CD4 >500: number analyzed (Participants) | 49 | 42
  Baseline CD4 >500 | 1522 [1178 to 1967] | 229 [145 to 359]
  Nadir CD4 <=350: number analyzed (Participants) | 40 | 37
  Nadir CD4 <=350 | 1390 [1040 to 1857] | 245 [151 to 395]
  Nadir CD4>350: number analyzed (Participants) | 32 | 27
  Nadir CD4>350 | 1752 [1303 to 2354] | 313 [186 to 528]

25. Secondary Outcome: Geometric Mean Titers for HPV 18 According to Participant Age, HIV Viral Load, CD4+ T Cell Count, and Nadir CD4 Level
Description: Geometric mean concentration of antibodies for HPV 18 at 7 and 24 months
Time Frame: at 7 and 24 Months
Population: Eligible participants who received at least one vaccination and who were sero-negative for HPV 18 at baseline with evaluable serum assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Month 7 Visit | Month 24 Visit
Number analyzed (Participants) | 88 | 73
mMU/mL
  Age<24 years: number analyzed (Participants) | 52 | 45
  Age<24 years | 310 [230 to 418] | 37 [25 to 55]
  Age>=24 years: number analyzed (Participants) | 36 | 28
  Age>=24 years | 281 [180 to 437] | 42 [26 to 69]
  Baseline HIV viral load <=75: number analyzed (Participants) | 78 | 64
  Baseline HIV viral load <=75 | 333 [258 to 431] | 42 [30 to 57]
  Baseline HIV viral load >75: number analyzed (Participants) | 10 | 9
  Baseline HIV viral load >75 | 123 [57 to 267] | 25 [7 to 86]
  Baseline CD4 <=500: number analyzed (Participants) | 33 | 28
  Baseline CD4 <=500 | 327 [209 to 511] | 45 [26 to 77]
  Baseline CD4 >500: number analyzed (Participants) | 55 | 45
  Baseline CD4 >500 | 282 [208 to 381] | 36 [25 to 52]
  Nadir CD4 <=350: number analyzed (Participants) | 52 | 44
  Nadir CD4 <=350 | 338 [240 to 476] | 42 [29 to 62]
  Nadir CD4>350: number analyzed (Participants) | 33 | 28
  Nadir CD4>350 | 268 [185 to 387] | 36 [21 to 62]

ADVERSE EVENTS:
Time Frame: From enrollment through 2 years after the first injection of Gardasil.
Description: All adverse events (AEs), regardless of severity, and whether or not ascribed to the study vaccine administration, were recorded. All Grade ≥ 2 laboratory values (except for CD4 cell counts) were recorded as AEs. After Week 32, only SAEs and AEs or symptoms > grade 3 or symptoms that were possibly, probably, or definitely related to the study vaccine were recorded. Subjects who were withdrawn from the study due to AEs were to be followed by the Investigator until the outcome was determined.
Arm/Group | Vaccination
All-Cause Mortality (participants affected / at risk) | 0/144
Serious Adverse Events (participants affected / at risk) | 5/144
Other Adverse Events (participants affected / at risk) | 59/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccination (N=144)
Skin infection (Infections and infestations) | 2 (2)
Gum infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Psychiatric disorders - other, specify (Psychiatric disorders) | 1 (1) — Homicidal ideation
Suicidal ideation (Psychiatric disorders) | 1 (3)
Suicide attempt (Psychiatric disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccination (N=144)
Diarrhea (Gastrointestinal disorders) | 8
Injection site reaction (General disorders) | 37
Neutrophil count decreased (Investigations) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Skin and subcutaneous tissue disorder - other, specify (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT01209325/Prot_SAP_001.pdf